CLINICAL TRIAL: NCT00005760
Title: A Pilot Study of the Metabolic Effects of Large Volume Liposuction in Overweight Women With Hyperinsulinemia, Impaired Glucose Tolerance and/or Type 2 Diabetes
Brief Title: Health Effects of Liposuction in Overweight Women With Elevated Insulin Levels, Impaired Glucose Tolerance and/or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000115; 00-CH-0115
Record Dates: First submitted 2000-05-26; First posted 2000-05-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Glucose Intolerance; Hyperinsulinemia; Diabetes Mellitus, Non Insulin Dependent; Obesity
Keywords: Dyslipidemia; Hypertension; Metabolic Syndrome X; Obesity; Subcutaneous Adipose Tissue; Visceral Abdominal Adipose Tissue
MeSH Terms: conditions — Glucose Intolerance; Hyperinsulinism; Diabetes Mellitus, Type 2; Obesity; Dyslipidemias; Hypertension; Metabolic Syndrome

SUMMARY:
This study is for women who have already decided to undergo liposuction at Georgetown University Medical Center in Washington, D.C. To take part in this study, a woman must first meet with the plastic surgeons there, and be accepted by them to have liposuction. This study will investigate whether large volume liposuction improves risk factors for heart disease in overweight women with type 2 (adult onset) diabetes, impaired glucose tolerance, or elevated blood insulin levels. Large volume liposuction is the surgical removal of at least 10 pounds (4.5 kg) of body fat, usually from the abdomen, hips or chest. Risk factors for heart disease include high blood pressure and elevated levels of blood lipids (cholesterol and triglycerides), blood glucose (sugar), and blood insulin. Subjects who participate in all parts of this study will receive a total of $930.00.

Overweight women 18 years or older with high blood insulin levels, impaired glucose tolerance, or type 2 diabetes, who are planning to have large volume liposuction performed at Georgetown University Medical Center in Washington, D.C., may be eligible for this study. For a subject to be accepted into this study, she must first meet with the plastic surgeons at Georgetown University Medical Center, and they have to agree to perform large volume liposuction. The decision that someone is suitable for liposuction is not under the control of the NIH or of any NIH investigator.

Those enrolled will undergo the following procedures at four separate times - before undergoing liposuction, 4 weeks after surgery, 4 months after surgery and 1 year after surgery:

* Body measurements - taken with calipers to measure several skinfold thicknesses (the width of a fat fold) and with a tape measure to measure the circumference of parts of the body.
* Urine sample and 6-hour urine collection - to test for pregnancy and to evaluate kidney function.
* Glucose tolerance test - measures insulin sensitivity and how the body uses sugar, how well insulin works, and insulin sensitivity. The procedure involves placement of two catheters (thin, flexible tubes) through a needle into a vein in each arm. Sugar water is infused into one catheter and 20 minutes into the test a small amount of insulin is injected. Blood samples are drawn from the other catheter at frequent intervals for a total of 5 hours.
* Electrocardiogram (ECG) and echocardiography - measure the heart's electrical activity and function.
* Abdominal computerized tomography (CT) scan - produces images for measuring body fat in the abdomen. (not done at the 4-week visit). Takes about half an hour to complete.
* DXA X-ray - measures body fat, muscle and bone mineral content. Takes about half an hour to complete.
* Bod Pod - capsule-like device used to determine the proportion of body weight composed of fat and non-fat tissue. Takes less than 10 minutes
* Bioelectric impedance analysis device - measures the proportions of body fat based on electrical conduction of a small electric current. Takes 2-3 minutes.
* 24-hour blood pressure monitoring - a device attached to a blood pressure cuff strapped to the arm measures blood pressure every 15 to 30 minutes continuously for 24 hours.
* Vascular reactivity tests - a blood pressure cuff is inflated for about 4 minutes before deflating, providing information on the function of the small blood vessels in the skin, as well as an idea of the function level of small blood vessels elsewhere in the body. Takes half an hour.
* Blood samples - collected to evaluate kidney and liver function and to measure body lipids, such as cholesterol, minerals, and other substances.

DETAILED DESCRIPTION:
Obesity is a major predisposing factor for future Type 2 diabetes because it is often associated with insulin resistance and impaired glucose tolerance. Insulin resistance has been suggested as the common link for other aspects of the cardiac dysmetabolic syndrome that includes hypertension, dyslipidemia, obesity, and macrovascular arterial disease. There are racial disparities in the prevalence of both obesity and Type 2 diabetes: Compared with non-Hispanic Caucasians, African American women have almost twice the prevalence of overweight, obesity, and Type 2 diabetes.

Because data from predominantly Caucasian populations suggest that the quantity of truncal (sometimes called upper body) adipose tissue, which includes the adipose tissue surrounding the abdominal viscera, is far more important for risk stratification than that found in the limbs or buttocks, which contain subcutaneous adipose tissue, it has been presumed that attempts at treatment of obesity should concentrate on reducing visceral fat. However, despite their greater risks for the complications of obesity, African Americans have less visceral abdominal adipose tissue than Caucasians matched for body weight. Further, recent metabolic studies suggest that upper body subcutaneous adipose tissue may play a significant role, particularly for African Americans, in the comorbid metabolic conditions associated with obesity.

With the advent of the large volume liposuction technique, selective removal of substantial quantities of subcutaneous adipose tissue has become possible. It is unknown whether the complications of obesity can be ameliorated by removal of subcutaneous adipose tissue, but one preliminary study suggests that fasting hyperinsulinism can be improved by this approach.

We propose to conduct a pilot study of 10 patients (five Caucasians and five African-Americans) who plan to undergo liposuction. We will investigate how large volume liposuction affects the metabolic complications of obesity in overweight patients who have hyperinsulinemia, impaired glucose tolerance, or type 2 diabetes. We will investigate the effects of liposuction on various indices of the cardiac dysmetabolic syndrome by performing studies of insulin sensitivity and lipid metabolism at four time points: before large volume liposuction, 1 month after liposuction, 4 months after liposuction, and 1 year after liposuction. At each visit we will study body composition, blood pressure, cardiac function, dietary habits, insulin insensitivity, free fatty acids, and lipid profiles.

ELIGIBILITY:
Patients must be in good general health. Patients with chronic stable complications of Type 2 diabetes or stable obesity related comorbid conditions will not be excluded.

Obesity: Defined as subjects having a body mass index greater than 30 kg/m(2). Weight must be less than 300 lb (136 kg) because of limits related to the DXA and CT scanners.

Patients with Type 2 Diabetes, impaired glucose tolerance, or hyperinsulinemia are eligible.

Patients' age must be greater than or equal to 18 years at the start of the study.

Patients must be planning to undergo large volume liposuction.

Premenopausal women participating in the study must have a negative pregnancy test at the start of the study and will be required to remain on some form of effective contraception for the duration of the study.

Patients recruited for the pilot study will be required to have all four grandparents and both parents to be either all non-Hispanic Caucasians or non-Hispanic African-American.

Volunteers with the presence of significant, unstable or evolving renal disease are not eligible. Subjects must not have calculated (age and weight corrected) creatinine clearances below 50 ml/min or significant worsening of serum creatinine levels during the course of the study (greater than 30% increase from baseline).

Volunteers with the presence of significant, unstable or evolving hepatic disease associated with SGOT and/or SGPT greater than 2.5 times normal are not eligible.

Volunteers with the presence of significant, evolving or unstable cardiac disease are not eligible. Subjects with NYHA stage 3 or 4 disease will be excluded from the study.

Volunteers with the presence of significant, evolving or unstable pulmonary disease including uncontrolled bronchial asthma and/or chronic bronchitis are not eligible.

Volunteers with the presence of other uncontrolled or unstable medical conditions including uncontrolled thyroid disease, Cushing's syndrome, autoimmune or gastrointestinal disease are not eligible.

Volunteers who are pregnant are not eligible.

Volunteers must not have uncontrolled Type 2 diabetes as evidenced by recent coma or pre-coma states, frequent episodes of hypoglycemia, predominantly severe hyperglycemia (plasma glucose greater than 400 mg/dl) in the past three months prior to study commencement, a glycosylated hemoglobin (HBA1C) value greater than 10 in the past three months prior to the study commencement, and frequent or recurrent episodes of ketosis (ketonuria and/or ketonemia).

Volunteers with uncontrolled, significant or evolving psychiatric/psychological syndromes which in the opinion of the investigators would place the patient at increased risk during the course of the study or would impede competence and/or ability to complete the study are not eligible.

Volunteers with current history of illicit substance abuse and/or alcoholism based on reported history and the CAGE questionnaire are not eligible.

Volunteers must not have a recent use (within the preceding 6 months) of anorexiant medications or medications that would affect nutrient absorption such as orlistat or acarbose.

Volunteers must not be receiving treatment with an insulin-sensitizing medication such as metformin or the thiazolidinediones. Use of insulin, meglitides or the sulphonylureas will not constitute an exclusion.

Volunteers with an absence of spontaneous menses for greater than 1 year are not eligible.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2000-05; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Pi-Sunyer FX, Laferrere B, Aronne LJ, Bray GA. Therapeutic controversy: Obesity--a modern-day epidemic. J Clin Endocrinol Metab. 1999 Jan;84(1):3-12. doi: 10.1210/jcem.84.1.5392-1. PMID 9920054
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Mokdad AH, Serdula MK, Dietz WH, Bowman BA, Marks JS, Koplan JP. The spread of the obesity epidemic in the United States, 1991-1998. JAMA. 1999 Oct 27;282(16):1519-22. doi: 10.1001/jama.282.16.1519. PMID 10546690